CLINICAL TRIAL: NCT01416961
Title: Phase I Study of High Linear Energy Transfer (Neutron) Therapy Followed by Concurrent Chemotherapy and Standard Photon Thoracic RT (TRT) in Stage III NSCLC (Non-Small Cell Lung Cancer) Patients
Brief Title: Integration of Neutron Therapy in the Treatment Plan for Stage III Non-Small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Neutron therapy has become unavailable
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Shirish Gadgeel, Physician Manager, Wayne State University Faculty; Associate Professor, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-005
Record Dates: First submitted 2011-08-10; First posted 2011-08-15 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Lung Cancer
Keywords: Squamous Cell; Non-squamous cell
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy; Cisplatin; Etoposide; etoposide phosphate; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Radiation Therapy — Concurrent chemo and photon radiation therapy will start within 7 days of completing neutron therapy. There will be a Day 1 of neutron therapy and a Day 1 of concurrent therapy.Photon radiation therapy will begin within 24 hours of the first cycle of chemotherapy and will be delivered 5 days per week, one fraction per day, in 1.8 Gy per fraction. High LET radiotherapy will be delivered in 1 NGy per fraction five days per week. High LET radiotherapy will be delivered first followed by combined chemoradiotherapy.
Drug: Chemotherapy - Squamous Cell Histologies — Cisplatin 50 mg/m2 administered on days 1,8, 29, 36; Etoposide 50 mg/m2 administered on days 1-5 and then again days 29-33
  Other Names: Platinol ®; Platinol®-AQ; CDDP; Toposar®; VePesid®; Etopophos®; VP-16; Etoposide phosphate
Drug: Chemotherapy - NSCLC other than squamous cell — Cisplatin 75 mg/m2 days 1,22,43; Pemetrexed 500 mg/m2 days 1,22,43
  Other Names: Alimta; Platinol ®; Platinol®-AQ; CDDP

SUMMARY:
This study is needed to assess the feasibility of integrating this therapy with current treatment regimens. If this study shows success a formal phase II test study to conduct feasibility will be the next step. The first dose level chosen for this study is 66Gy of radiation to the tumor between LET and standard photon therapy. This dose is the current standard of care for stage III . If this dose is found to be feasible then the dose of LET will escalate to the total dose of 74Gy.

ELIGIBILITY:
Inclusion Criteria:

* IIIA :

Histologic or cytologic diagnosis of ipsilateral mediastinal lymph node involvement, or Tumors greater than 7 cm or with chest wall invasion, or involvement of one of the following diaphragm, phrenic nerve, mediastinal pleura or parietal pericardium with hilar or mediastinal lymph node involvement.

More than one mediastinal lymph node enlarged on CT scan and the same lymph nodes positive on PET scans or Paralyzed left vocal cord with separate lung primary distinct from the aorto-pulmonary lymph nodes on the CT scan.

Evidence of tumor extension into the mediastinum and/or mediastinal structures either at the time of mediastinoscopy, bronchoscopy or on CT scans.

* IIIB:

Histologic or cytologic diagnosis of N3 lymph node involvement; or Enlarged N3 lymph nodes on CT scan that are positive on PET scan as well. Patient must not have extension of lymph node involvement to cervical lymph nodes other than supraclavicular lymph nodes; or Right sided primary with left vocal cord paralysis; or Patients with a nodules in the same lung but no other areas of involvement. Patients with prior surgically resected stage I NSCLC who did not receive any adjuvant therapy, who now have stage IIIA or B NSCLC will be eligible.

* Age ≥ 18 years
* SWOG performance status 0 or 1 (see Appendix)
* Adequate organ function as evidenced by Absolute neutrophil count of ≥ 1.5 x 10(9)/L, Platelet count ≥ 100,000 x 109/L Serum creatinine ≤ 1.5 times the institutional upper limit of normal (ULN), Calculated creatinine clearance (Cockcroft-Gault formula) of ≥ 45mL/min, Serum bilirubin ≤ ULN, Transaminases (SGOT and/or SGPT) ≤ 1.5 times institutional ULN and alkaline phosphatase ≤ 2.5 times ULN, FEV1 of ≥ 1 liter and DLCO > 50% of predicted.
* Patient should undergo brain imaging (CT scan or MRI) to rule out brain metastases.
* Signed informed consent that details the investigational nature of the study according to institutional and federal guidelines.
* Registered with Clinical Trials Office at Karmanos Cancer Institute/Wayne State University.

Exclusion Criteria:

* Prior chemotherapy, radiation for any malignancy in which they received any thoracic radiotherapy.
* Patients with concurrent malignancy. Patients with prior or concurrent malignancy will be allowed as long as the treating physician considers it unlikely to impact the clinical outcome of the patient.
* Patients with peripheral neuropathy ≥ 2.
* Serious medical illness including but not limited to uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction or cerebrovascular event with 6 months of registration, history of chronic active hepatitis or history of HIV or an active bacterial infection will not be eligible.
* Inability or unwillingness to take folic acid or Vitamin B12 or dexamethasone.
* Pregnant or lactating women. All pre-menopausal and peri-menopausal women should have a urine test for pregnancy within a week of starting therapy. All patients of child bearing potential should agree to use an effective contraceptive method.
* Patients should not participate in any other therapeutic investigational study while taking part in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assess Dose levels (DLT & MTD)integrating 2 dose levels of neutron tx in 2 diff regimens of approx 12 pts/trt; If 1st dose level feasible but not 2nd dose level in either cohorts then 12 pts will be trted at 1st dose level for that particular cohort | up to one month after therapy
  Lab value chgs (CBC w/diff, electrolytes, serum cr., calc. cr. clearance, bilirubin, AST, ALT, ca, mg, LDH, albumin)& for AE's-wks. 2, 5, 6, 8 & 1 mth. after therapy. Dose Limiting Toxicities (DLT): Gr 3/4 non-hematologic tox that is trtment related; Gr 4 thrombocytopenia, Gr 3/4 neutropenic fever or gr 4 neutropenia lasting > 7 days. Assess 2 dose levels, the maximum tolerated dose (MTD) of neutron therapy-dose at which < 33% of the pts. experience DLT.

SECONDARY OUTCOMES:
To assess the Progression Free Survival (PFS), and response rate in these patients. | CT scan of the chest to assess the status of the cancer within 30 days of completion of therapy. If the patient has had complete or partial response, then a repeat scan no sooner than 4 weeks should be done to confirm the response.
To assess the expression of p16 expression, ERCC1 and TS expression in tumors of enrolled patients and assess the correlation of these markers with response rate and progression free survival. | Archival tissue samples collected at baseline will be assessed at baseline & 1 month after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M. Gadgeel, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute